CLINICAL TRIAL: NCT04470830
Title: Post-Marketing Surveillance (Usage Results Study) of Azilsartan Medoxomil/Chlorthalidone FDC in the Treatment of Patients With Essential Hypertension in South Korea
Brief Title: A Study for PMS of AZL-M/CLD FDC in the Treatment of Participants With Essential HTN in South Korea
Status: Completed | Type: Observational
Sponsor: Celltrion Pharm, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-491-5001; U1111-1252-3527 (Registry Identifier: WHO)
Record Dates: First submitted 2020-07-13; First posted 2020-07-14 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Essential Hypertension
Keywords: Drug Therapy
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With Essential Hypertension: Participants diagnosed with essential hypertension who have been treated with azilsartan medoxomil/chlorthalidone FDC as an early therapy for participants whose blood pressure is not properly controlled by monotherapy or who require administration of multiple drugs in order to reach the target blood pressure, will be observed prospectively over a period of 5 years.

SUMMARY:
The purpose of this study is to evaluate the safety by assessing all serious and non-serious adverse events (AEs), irrespective of relatedness or expectedness, as well as other safety parameters including laboratory values, serious adverse events (SAEs)/serious adverse drug reactions (ADRs), unexpected AEs and ADRs that are not reflected on the precaution in the use, ADRs already known, non-serious ADRs and other safety related information (laboratory values changes, etc).

DETAILED DESCRIPTION:
This is a long-term prospective, observational post-marketing surveillance study of azilsartan medoxomil/chlorthalidone FDC in participants with essential hypertension. The study will assess the safety and effectiveness of azilsartan medoxomil/chlorthalidone FDC prescribed as a monotherapy or taken concomitantly with other anti-hypertension therapies in participants whose blood pressure is not properly controlled by azilsartan medoxomil monotherapy or who require administration of multiple drugs in order to reach the target blood pressure in routine clinical settings.

The study will enroll and will consider approximately 600 participants. These participants will be grouped with the ones treated with azilsartan medoximil monotherpy. The data will be prospectively collected, at the centers from medical files and recorded into electronic case report forms (e-CRFs). All the participants will be assigned to a single observational cohort:

• Participants With Essential Hypertension

The multi-center study will be conducted in South Korea. Data collection will be based on routinely scheduled and emergency visits over the surveillance period, scheduled at Visit 1 (Baseline), Visit 2 (6 weeks), Visit 3 (at least 3 months to 6 months) and Visit 4 (6 months or more up to 9 months) after drug administration. The overall duration of the study will be approximately 5 years. All participants will be followed up for 9 months after drug administration.

ELIGIBILITY:
Inclusion Criteria:

1. Has a SBP or DBP >=140 or 90 mmHg, respectively.
2. Newly prescribed azilsartan medoxomil/chlorthalidone FDC as an early therapy for participants whose blood pressure is not properly controlled by monotherapy with azilsartan medoxomil or who require administration of multiple drugs in order to reach the target blood pressure in participants with stage 2 hypertension.

Exclusion Criteria:

1. With anuria.
2. With refractory hypokalemia.
3. With severe hepatic or renal impairment (estimate glomerular filtration rate [eGFR] <30 milliliter per minute per 1.73 square meter [mL/min/1.73 m^2]).
4. With hyponatremia, hypercalcemia.
5. With symptomatic hyperuricemia (history of gout and urate stone).
6. With untreated Addison's disease.
7. Receiving lithium therapy.
8. Administrating terfenadine and/or astemizole.
9. Use of aliskiren in combination with study drug in participants with diabetes or with moderate to severe renal impairment (glomerular filtration rate [GFR] <60 mL/min/1.73m^2).
10. Participating in a clinical trial evaluating a hypertension treatment.
11. Treated with azilsartan medoxomil / chlorthalidone FDC outside of the locally approved label in South Korea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have administered azilsartan medoxomil/chlorthalidone FDC as an early therapy for participants whose blood pressure is not properly controlled by monotherapy or who require administration of multiple drugs in order to reach the target blood pressure will be observed prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 718 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants who Experience at Least one AE and SAE | Baseline up to Month 9

SECONDARY OUTCOMES:
Change From Baseline in Blood Pressure Including Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) | Baseline up to Month 9
  Blood pressure (SBP and DBP) will be measured in millimeter of mercury (mmHg).
Percentage of Participants who Achieve Clinic DBP less than (<) 90 mmHg and/or reduction of Greater than or equal to (>=) 10 mmHg | Baseline up to Month 9
Percentage of Participants who Achieve Clinic SBP <140 mmHg and/or reduction of >=20 mmHg | Baseline up to Month 9
Percentage of Participants who Achieve Both Clinic DBP <90 mmHg and/or Reduction of >=10 mmHg and Clinic SBP <140 mmHg and/or Reduction of >=20 mmHg | Baseline up to Month 9
Change From Baseline in Serum Creatinine Level, Serum Uric Acid Level and Serum Lipid Profile | Baseline up to Month 9
  Serum creatinine level, serum uric acid level, and serum lipid profile will be measured in milligram per deciliter (mg/dL).
Change From Baseline in Blood Potassium Level | Baseline up to Month 9
  Blood potassium level will be measured in millimole per liter (mmol/L).
Change From Baseline in Blood Sodium Profiles | Baseline up to Month 9
  Blood sodium profiles will be measured in milliequivalent per liter (mEq/L).
Final Effectiveness Rate as Assessed by the Investigator | Baseline up to Month 9
  Effectiveness rate: percentage of participants who achieved effectiveness over total number of assessable effectiveness analysis population, and is calculated as number of effective participants/total number of participants in group, multiplied by 100. Final effectiveness will be assessed based on: Improved (symptoms have improved or it is considered to have had a maintenance effect); Unchanged (no significant change from pre-administration, not considered to have had a maintenance effect); Worsened (symptoms have worsened compared to pre-administration); Unassessable (unable to assess due to grounds such as missing effectiveness variables, follow up loss, etc.). Maintenance effect: cases where the likelihood of worsened symptoms is high with discontinuation of medication, or equivalent effect to existing drugs is sustained when substituted with existing drugs. Effectiveness rate is determined by classifying 'Improved' as "Effective" and 'Unchanged' and 'Worsened' as "Ineffective".

CONTACTS AND LOCATIONS:
Locations (1):
- Yeungnam University Medical Center, Daegu, Gyeongsangbuk-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.